CLINICAL TRIAL: NCT07089264
Title: Physical Rehabilitation in Patients With Complex Congenital Heart Disease
Acronym: Rehabkids
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025physicalrehab; CAAE 22130219.0.0000.0060 (Other: CEP - FMUSP)
Record Dates: First submitted 2025-06-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: congenital heart disease; quality of life; cardiopulmonary; six-minute walk test; physical rehabilitation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: This cross-sectional study included 15 children with complex congenital heart disease who underwent surgical correction. Different examinations were performed: cardiopulmonary exercise was used; and the six-minute walk test (6MWT) was used to determine functional capacity, the Peds - QL cardiac version questionnaire was used to determine quality of life. Descriptive analysis of patients was performed for all the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Rehabilitation (Other): Physical Rehabilitation in 36 sessions
  Interventions: Other: Physical rehabilitation

INTERVENTIONS:
Other: Physical rehabilitation — Physical Rehabilitation in 36 sessions

SUMMARY:
Studies have shown that patients with congenital heart disease have functional changes compared to healthy individuals. Several interventions can be performed to minimize these changes; physical rehabilitation is one of these possible treatments that can generate numerous benefits for patients. The aim of this study is to evaluate the response to physical rehabilitation in patients after surgical correction of congenital heart disease.

Methods This cross-sectional study included patients with complex congenital heart disease who underwent surgical correction. Different examinations were performed: cardiopulmonary exercise was used; and the six-minute walk test was used to determine functional capacity, the quality of life cardiac version questionnaire was used to determine quality of life. Descriptive analysis of patients was performed for all the data.

DETAILED DESCRIPTION:
Study design and population This cross-sectional study analyzed those patients with complex congenital heart disease who underwent surgical correction at Hospital do Coração, São Paulo - Brazil. The institutional ethics committees on human research approved . All the subjects signed consent forms before starting the protocol.

The survey of patients eligible for the physical rehabilitation protocol was conducted at the Congenital Cardiology Outpatient Clinic of the Hospital do Coração. Patients currently under clinical follow-up the investigators selected for inclusion in the study. The protocol was presented to the medical team, and patients who did not exhibit neuromuscular, pulmonary, or complex orthopedic conditions that could interfere with the performance of the assessments the investigators chosen.

Transthoracic echocardiography The transthoracic echocardiographic evaluation will be performed using the two-dimensional technique, always by an echocardiographer. All images will be obtained by software, using an appropriate transducer. Echocardiographic measurements will be made in accordance with the recommendations of the congenital heart disease consensus.

Cardiopulmonary exercise test The cardiopulmonary exercise test was performed using a treadmill exercise test equipped with a metabolic analyzer. This assessment aimed to determine the subject's maximal cardiopulmonary capacity.

Blood pressure measurements were taken at rest, every two minutes during exercise, and every minute during the recovery phase. All readings were taken by the same observer, using the auscultatory method to ensure consistency.

A customized ramp-up protocol based on the modified Balke approach was employed, featuring an increase in speed during the first 3 minutes, followed by a two percent rise increase in incline every minute until the participant reached exhaustion.

Ventilation, oxygen consumption, and carbon dioxide production were assessed using a breath-by-breath analysis technique, from which ventilatory thresholds were calculated. Maximal functional capacity was determined using absolute peak oxygen and relative peak oxygen, expressed as a percentage of predicted values for age- and sex-matched healthy individuals.

Additional parameters, including the oxygen uptake efficiency slope and the ventilatory equivalent for carbon dioxide, were also measured and analyzed.

Six-minute walk test A submaximal analysis of physical capacity was conducted using the six-minute walk test, following the protocol.

The patients were instructed to walk as quickly as possible without running for six minutes, while the distance covered was recorded. Breaks during the walk were allowed if needed. The data analyzed included the distance covered in meters, heart rate, respiratory rate, peripheral oxygen saturation, blood pressure, and the fatigue. These measurements were taken at rest one minute before the test, immediately after the test, two minutes after the test if there was an interruption, and five minutes after the test.

Quality of life To evaluate quality of life, the investigators employed the Pediatric Quality of Life Inventory cardiac version questionnaire. This instrument encompasses various domains, including symptoms, treatment, physical appearance, anxiety related to treatment, challenges with understanding and communication. The questionnaire is completed by both the patient and their parents.

ELIGIBILITY:
Inclusion Criteria:

* no previous or current history of other non-cardiological disease
* patients undergoing complex congenital heart surgeries with a minimum postoperative period of 1 year
* clinically stable; with no complex arrhythmia(s) in the last electrocardiogram or clinical evaluation
* with medical monitoring
* clinical clearance to carry out the protocols
* consent with the Free and Informed Consent Form (FICF) and Assent Form signed by the guardian and the patient respectively.

Exclusion Criteria:

* patients with musculoskeletal or neuropsychiatric alterations without the possibility of performing a functional test (ergospirometry test),
* hemodynamically unstable patients
* severe respiratory or metabolic conditions
* patients residing in regions far from São Paulo,
* patients which make frequent visits to the institution unfeasible
* patients who do not attend the rehabilitation program or those for whom it was not possible to maintain and update registration data.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the response to aerobic activity and peripheral muscle strength training in children with congenital heart disease. | In 36 physical rehabilitation sessions, twice a week lasting about 4.5 weeks
  Quantify the speed (which is the measurement of distance in kilometers divided by time in hours) of walking and running in km/h during aerobic exercises on a treadmill; evaluate the load capacity in kilograms in lower and upper limb exercises.

SECONDARY OUTCOMES:
Quality of life assessment | The test lasts approximately 10 minutes and will be performed on day 1 of care and on the last day - day 36.
  To assess quality of life, we used the Pediatric Quality of Life Inventory (PedsQL) questionnaire, cardiac version. This instrument covers several domains such as: symptoms, treatment, physical appearance, anxiety related to treatment and difficulties in understanding and communication. The questionnaire is completed by both the patient and their parents. These questions are presented in which the highest score (100) represents the best quality of life and the lowest score (0) represents the worst quality of life.
The cardiopulmonary test - ergospirometry | The test lasts approximately 30 minutes and will be performed on the first day - day 1 of care and on the last day - day 36 of care for discharge.
  The test was performed using an individualized ramp protocol on a treadmill, monitored by 12-lead electrocardiogram, heart rate in beats per minute (bpm), and blood pressure in millimeters of mercury (mmHg) using the digital method. The metabolic analyzer and exhaled gas collection during the rest, exercise, and recovery phases were performed using a mask connected to a gas analysis system, calibrated before each test. Direct measurements of minute ventilation in liters (L), peak oxygen consumption in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min), and carbon dioxide output as the partial pressure of carbon dioxide (PaCO2) were performed.
Submaximal exercise test - six-minute walk test | The test lasts approximately 10 minutes and will be performed on day 1 of care and on the last day - day 36.
  A submaximal analysis of physical capacity was conducted using the six-minute walk test (6MWT), following the protocol of the American Thoracic Society. The patients were instructed to walk as quickly as possible without running for six minutes, while the distance covered was recorded. Breaks during the walk were allowed if needed. The data analyzed included the distance covered in meters, heart rate, respiratory rate, peripheral oxygen saturation, blood pressure, and the Modified Borg Scale for Fatigue. These measurements were taken at rest one minute before the test, immediately after the test, two minutes after the test if there was an interruption, and five minutes after the test
Assessment of cardiac function | The test lasts approximately 30 minutes and will be performed on the first day - day 1 of care and on the last day - day 36 of care for discharge.
  Transthoracic echocardiographic assessment will be performed using the two-dimensional technique. Echocardiographic measurements will be made in accordance with the recommendations of the American Society of Echocardiography and the Congenital Heart Disease Consensus.
  The assessment of atrioventricular valve function will be made based on the degree of stenosis through analysis of the mean diastolic gradient measured in millimeters of mercury (mmHg) and the assessment of the degree of regurgitation through color Doppler to identify the direction and extent of reverse blood flow. The severity of regurgitation can be classified as mild, moderate or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Coração, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
If any researcher is interested in replicating the study, please contact us for further clarification.
Supporting Information: Study Protocol
Time Frame: If any researcher is interested in replicating the study, please contact us for further clarification.
Access Criteria: If any researcher is interested in replicating the study, please contact us for further clarification.

REFERENCES:
- [Background] Silveira JBPDM, Turquetto ALR, Amato LP, Agostinho DR, Caneo LF, Binotto MA, da Costa Soares Lopes MI, Rodrigues JC, Santos MVB, Oliveira PA, TanaKa ACS, Jatene MB. Comparative Analysis of Respiratory and Functional Outcomes in Children Post-Fontan Procedure Versus Healthy Peers. Pediatr Cardiol. 2025 Dec;46(8):2379-2390. doi: 10.1007/s00246-024-03666-8. Epub 2024 Oct 21. PMID 39432096